CLINICAL TRIAL: NCT02370173
Title: A Non-Pharmacological Method for Enhancing Sleep in PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Principal Investigator, William D. Killgore, Principal Investigator, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1407389306A003
Record Dates: First submitted 2014-10-15; First posted 2015-02-24 (Estimated); Results first posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: PTSD; Sleep Problems
Keywords: PTSD; Stress; Sleep Problems; Brain imaging; fMRI
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTSD wavelength-1 bright light (Experimental): 30 minutes of daily light exposure for 6 weeks
  Interventions: Device: PTSD wavelength-1 bright light
- PTSD wavelength-2 bright light (Placebo Comparator): 30 minutes of daily light exposure for 6 weeks
  Interventions: Device: PTSD wavelength-2 bright light

INTERVENTIONS:
Device: PTSD wavelength-1 bright light — 6 weeks of daily light exposure, 30 minutes per morning.
  Arms: PTSD wavelength-1 bright light
Device: PTSD wavelength-2 bright light — 6 weeks daily light exposure, 30 minutes per morning.
  Arms: PTSD wavelength-2 bright light

SUMMARY:
Sleep disturbance is nearly ubiquitous among individuals suffering from PTSD and is a major problem among service members returning from combat deployments. The proposed study aims to test a novel, inexpensive, and easy to use approach to improving sleep among service members with PTSD.

Primary outcome measures will include not only PTSD symptom improvement but also include neuroimaging of brain structure, function, connectivity, and neurochemistry changes. The proposal is firmly grounded in the emerging scientific literature regarding sleep, light exposure, brain function, anxiety, and resilience. Prior evidence suggests that bright light therapy is effective for improving mood and fatigue, and our pilot data further suggest that this treatment may be effective for improving daytime sleepiness and brain functioning in brain injured individuals. Thus, this intervention, in our own research and in the work of others, has been shown to affect critical sleep regulatory systems. Improving sleep may be a vital component of recovery in these service members. Our approach would directly address this issue. Our preliminary data have shown that this approach is extremely well tolerated and is effective for improving sleep, mood, cognitive performance, and brain function among individuals with brain injuries.

Finally, the potential impact of this study is high because of the capability of transitioning the research to direct clinical application almost immediately. If the bright light treatment is demonstrated as effective, this approach would be readily available for nearly immediate large-scale implementation, as the devices have been widely used for years in other contexts, are already safety tested, and commercially available from several manufacturers for a very low cost. Thus, the impact of this research on treating PTSD would be high and immediate.

ELIGIBILITY:
* Having experienced a traumatic event within the past 10 years
* Right handedness
* 18-50 years old
* Primary language is English
* No metal in body

Further eligibility will be determined through a phone screening. Please call (520) 626-8591 or go to uascanlab.com to check your eligibility for this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2014-09; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Killgore, Ph.D., Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Psychiatry Department, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PTSD Wavelength-1 Amber: 30 minutes of daily light exposure for 6 weeks
  PTSD wavelength-1 bright light: 6 weeks of daily light exposure, 30 minutes per morning.
- PTSD Wavelength-2 Blue: 30 minutes of daily light exposure for 6 weeks
  PTSD wavelength-2 bright light: 6 weeks daily light exposure, 30 minutes per morning.
Period: Overall Study
Arm/Group | PTSD Wavelength-1 Amber | PTSD Wavelength-2 Blue
Started | 43 | 47
Completed | 40 | 44
Not Completed | 3 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTSD Wavelength-1 Amber | PTSD Wavelength-2 Blue | Total
Number analyzed (Participants) | 43 | 47 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 47 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.07 (8.39) | 32.02 (8.99) | 31.38 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 29 | 31 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 31 | 59
  Hispanic/Latino | 8 | 9 | 17
  Black/African American | 2 | 2 | 4
  Asian/Pacific Islander | 0 | 1 | 1
  Other | 2 | 4 | 6
  Native American/American Indian | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 43 | 47 | 90

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency
Description: Actigraphy was used as a measurement of individual sleep efficiency calculating total sleep time (minutes asleep) divided by total rest time (time in bed- minutes in bed). This produces a percentage efficiency calculation that can range 0-100%, higher percentages indicates more time asleep while in bed.
Time Frame: Sleep Efficiency was calculated at Baseline (Pre-Treatment) and Post-Treatment (6 Weeks after Baseline)
Population: Because the rows in the outcome measure data table correspond to different timepoints, and because in some cases, data from certain measures were unusable, the number of individuals analyzed at each timepoint differs from the overall number analyzed (i.e. the number of unique individuals whose data were factored into the below descriptive statistics).
Measure: Mean (Standard Deviation); unit: Percentage of Sleep
Arm/Group | PTSD Wavelength-1 Bright Light | PTSD Wavelength-2 Bright Light
Number analyzed (Participants) | 40 | 44
Percentage of Sleep
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 88.13 (3.96) | 89.95 (3.17)
  Post-Treatment: number analyzed (Participants) | 36 | 43
  Post-Treatment | 89.31 (3.58) | 89.20 (4.03)

2. Primary Outcome: Subjective Sleep Quality
Description: Pittsburgh Sleep Quality Index is a measurement of subjective self-report sleep quality that uses both free response and Likert scale responses. The range of scores possible are 0 to 21. Higher scores indicate worse subjective sleep quality.
Time Frame: Results 6 weeks post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTSD Wavelength-1 Amber | PTSD Wavelength-2 Blue
Number analyzed (Participants) | 38 | 44
score on a scale
  Baseline: number analyzed (Participants) | 36 | 43
  Baseline | 9.08 (3.42) | 9.86 (3.01)
  Post-Treatment | 7.53 (3.12) | 8.34 (3.24)

3. Primary Outcome: Neural Activation During Functional Magnetic Resonance Imaging (fMRI) Emotion Processing Task
Description: Activation of medial prefrontal cortex and anterior cingulate cortex (also prefrontal) during functional magnetic resonance imaging (fMRI) Backward Masked Affect Task (BMAT) emotion processing task. Contrast weight/effect scores for prefrontal area [MNI coordinates: 18,42,12] measured contrasts in activation between neutral images and activation when emotional images (fear images) were presented during the task. Higher scores indicate a greater difference or contrast between the neutral signal and emotional signal during the fMRI task.
Time Frame: Baseline (Pre-Treatment) and Post-Treatment (6 Weeks after Baseline)
Measure: Mean (Standard Error); unit: Arbitrary units
Arm/Group | PTSD Wavelength-1 Amber | PTSD Wavelength-2 Blue
Number analyzed (Participants) | 40 | 44
Arbitrary units
  Baseline | 0.0158 (0.0213) | -0.0843 (0.0248)
  Post-Treatment | 0.0445 (0.0242) | 0.0857 (0.0234)

4. Primary Outcome: Performance on Neuropsychological Assessment
Description: The Repeatable Battery for the Assessment of Neuropsychological Status will be utilized to measure overall neurocognitive performance. It covers five domains of cognition: Immediate Memory, Visuospatial/Constructional, Language, Attention, and Delayed Memory resulting in a total neurocognitive performance score. The range of overall total neurocognitive performance scores is 40-160 points. Higher scores on this scale represent a higher capacity for executive function.
Time Frame: Performance results at 6 weeks post-treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | PTSD Wavelength-1 Bright Light | PTSD Wavelength-2 Bright Light
Number analyzed (Participants) | 40 | 44
Points
  Baseline | 89.95 (12.46) | 93.16 (12.46)
  Post-Treatment: number analyzed (Participants) | 38 | 43
  Post-Treatment | 91.40 (13.40) | 95.42 (14.30)

5. Primary Outcome: PTSD Symptoms
Description: Post Traumatic Stress Disorder Checklist 5 (PCL-5).The PTSD Checklist for DSM-5 is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. Items are summed to provide a total severity score (range = 0-80). Higher scores indicate greater presence or severity of PTSD symptoms.
Time Frame: Performance results at 6 weeks post-treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTSD Wavelength-1 Bright Light | PTSD Wavelength-2 Bright Light
Number analyzed (Participants) | 40 | 44
score on a scale
  Baseline | 12.58 (3.5) | 13 (2.91)
  Post Treatment | 7.84 (4.40) | 9.02 (4.55)

6. Primary Outcome: Daytime Sleepiness (ESS)
Description: Epworth Sleepiness Scale is a subjective measure of daytime sleepiness. This is on a 4-point Likert scale, each item has a range of 0 to 3 points. The total score range for this is 0-24 points. Higher scores indicate more severe daytime sleepiness.
Time Frame: Performance results at 6 weeks post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTSD Wavelength-1 Bright Light | PTSD Wavelength-2 Bright Light
Number analyzed (Participants) | 40 | 44
score on a scale
  Baseline: number analyzed (Participants) | 40 | 43
  Baseline | 9.93 (4.46) | 9.61 (4.05)
  Post-Treatment: number analyzed (Participants) | 38 | 44
  Post-Treatment | 8.82 (4.13) | 8.82 (3.77)

7. Primary Outcome: Daytime Sleepiness (SSS)
Description: Stanford Sleepiness Scale is a one item scale assessing current level of alertness. The range of points possible is 1-7, with higher scores indicating that sleep onset is soon. This scale was given at three different time points during baseline assessment and post treatment.
Time Frame: Performance results at 6 weeks post-treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTSD Wavelength-1 Bright Light | PTSD Wavelength-2 Bright Light
Number analyzed (Participants) | 40 | 44
units on a scale
  Baseline - Administration 1 | 3.57 (1.48) | 3.80 (1.32)
  Baseline - Administration 2 | 3.60 (1.38) | 3.75 (1.31)
  Baseline - Administration 3 | 3.38 (1.409) | 3.30 (1.13)
  Post-Treatment - Administration 1 | 3.47 (1.34) | 3.49 (1.39)
  Post-Treatment - Administration 2 | 3.79 (1.30) | 3.35 (1.93)
  Post-Treatment - Administration 3 | 3 (1.13) | 2.93 (1.26)

8. Primary Outcome: Daytime Sleepiness (MSLT)
Description: Multiple Sleep Latency Test (MSLT). Participants were administered a modified Multiple Sleep Latency Test. In the multiple sleep latency test (MSLT), the participant was given 3 opportunities to nap for 20 minutes every two hours. Sleep latency scores are calculated in the number of seconds to fall asleep during their mandated sleep session. Range is from 0 seconds to 1200 seconds.
Time Frame: Change from baseline performance at 6 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PTSD Wavelength-1 Bright Light | PTSD Wavelength-2 Bright Light
Number analyzed (Participants) | 38 | 43
seconds
  Mean Sleep Latency in Seconds For First Administered Nap at Baseline Visit | 486.84 (359.27) | 487.67 (365.97)
  Mean Sleep Latency in Seconds For Second Administered Nap at Baseline Visit | 334.05 (271.12) | 390 (347.79)
  Mean Sleep Latency in Seconds For Third Administered Nap at Baseline Visit | 489.20 (411.4) | 520.71 (408.65)
  Mean Sleep Latency in Seconds For First Administered Nap while receiving Bright Light | 597.63 (459.83) | 552.75 (420.65)
  Mean Sleep Latency in Seconds For Second Administered Nap while receiving Bright Light | 481.67 (400.82) | 454.74 (405.23)
  Mean Sleep Latency in Seconds For Third Administered Nap while receiving Bright Light | 630.00 (498.96) | 494.62 (382.76)

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | PTSD Wavelength-1 Amber | PTSD Wavelength-2 Blue
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/47
Other Adverse Events (participants affected / at risk) | 0/43 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT02370173/Prot_SAP_000.pdf